CLINICAL TRIAL: NCT06610019
Title: Risk Stratification of Ischemic and Non-ischemic Cardiomyopathies in Racial and Ethnic Minority Groups in the Bronx - Cardiovascular Multimodality Imaging Study
Brief Title: Cardiovascular Multimodality Imaging Study
Status: Recruiting | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-14552
Record Dates: First submitted 2024-09-18; First posted 2024-09-24 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Non-ischemic Cardiomyopathy; Cardiomyopathies; Hypertrophic Cardiomyopathy; Right Ventricular Arrhythmogenic Cardiomyopathy; Cardiac Amyloidosis; Anderson Fabry Disease; Sarcoidosis; Cancer Therapy-related Cardiac Dysfunction; Ventricular Arrythmia; Heart Failure
Keywords: Cardiovascular Mortalities; Cardiomagnetic Resonance (CMR) Imaging; Prospective
MeSH Terms: conditions — Cardiomyopathies; Cardiomyopathy, Hypertrophic; Arrhythmogenic Right Ventricular Dysplasia; Amyloid Neuropathies, Familial; Fabry Disease; Sarcoidosis; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Determining the etiology of cardiomyopathy is of high clinical importance for optimal treatment strategy and prediction of prognosis. There is increased risk for cardiovascular disease and higher propensity for cardiovascular related mortality among Black and non-Hispanic White patients. Recently, advanced cardiac imaging has become a vital tool in diagnosis and risk stratification of cardiovascular disease. Very limited data is available on the prevalence and characteristics of different cardiovascular diseases in Hispanic and African American minority groups, therefore, studying different racial and ethnic minority groups in the Bronx population is an exceptionally valuable source to determine the prevalence of cardiomyopathies among minority groups along with study survival in this population. This study aims to determine the etiology of cardiovascular disease in a diverse patient population by utilizing various cardiovascular imaging modalities, with a focus on cardiac magnetic resonance (CMR) imaging and to develop risk stratification models by applying advanced cardiovascular imaging markers.

DETAILED DESCRIPTION:
Significant Hispanic and African American populations live in the Bronx and belong to the Montefiore Health System. Based on literature data, African Americans and Hispanics have a higher incidence of morbidity and mortality for various cardiovascular diseases (CVD) compared to non-Hispanic Whites. More than 53 million Hispanics currently live in the United States, which is 17% of the total US population and is expected to constitute 30% of the total US population by 2050. The increased risk for CVD is also well documented in the African American minority group. Although limited data is available on the prevalence and characteristics of different cardiovascular diseases in these minority groups. During the last two decades, advanced cardiovascular imaging modalities such as cardiovascular magnetic resonance (CMR) imaging became trusted tools in the risk stratification of patients with ischemic and non-ischemic cardiomyopathies.

Cardiovascular magnetic resonance (CMR) imaging is the gold standard for quantifying chamber size and function. In addition to ejection fraction, CMR feature-tracking (CMR-FT) is a new postprocessing technique that allows the assessment of myocardial mechanics from routinely acquired cine images without specialized additional pulse sequences. Basic global longitudinal strain has been proved as a predictive marker in non-ischemic cardiomyopathy (NICM). CMR imaging can also provide tissue-specific information about the myocardium using specific techniques such as late gadolinium enhancement (LGE) or other quantitative parameters like T1 mapping, both native and with measurement of extracellular volume fraction. Based on this, CMR imaging is an optimal modality to differentiate ischemic cardiomyopathy (ICM) and non-ischemic myocardial disease and diagnose different forms of NICM.

NICM represents a heterogeneous group of patients with multiple underlying etiologies. The pathogenesis of NICM with ventricular dilatation and reduced cardiac function in the absence of flow-limiting coronary artery disease (CAD) can be genetic, inflammatory, toxic, or viral. However, in the vast majority of cases, the origin is unclear. NICM may be either primary e.g. Hypertrophic cardiomyopathy (HCM), Right ventricular Arrhythmogenic Cardiomyopathy (ARVC), or secondary to systemic diseases such as Cardiac amyloidosis (CA), Anderson-Fabry disease, Sarcoidosis, or even iatrogenic as Cancer therapy-related cardiac dysfunction (CTRCD). Determining the etiology of cardiomyopathy is of high clinical importance for optimal treatment strategy and prediction of prognosis.

Upon further review, the Einstein Institutional Review Board (IRB) has determined that this is an ongoing, retrospective registry. and that there is no prospective component.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient (18 years or older) referred for a cardiovascular magnetic resonance (CMR) imaging study in the Montefiore Health System

Exclusion Criteria:

* Any patient who does not meet above criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients who receive a CMR study within the Montefiore Health System.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | From index CMR imaging to time of chart review, up to 5 years
  The number of patients who died from any cause will be summarized and reported using basic descriptive statistics.
Sudden Cardiac Death | From index CMR imaging to time of chart review, up to 5 years
  The number of patients who died from any cardiovascular-specific mortality will be summarized and reported using basic descriptive statistics.

SECONDARY OUTCOMES:
Heart Failure Hospitalizations | From index CMR imaging to time of chart review, up to 5 years
  The number of patients hospitalized with a primary diagnosis of heart failure will be summarized and reported using basic descriptive statistics.
Total Hospitalizations | From index CMR imaging to time of chart review, up to 5 years
  The number of patients hospitalized with any diagnosis will be summarized and reported using basic descriptive statistics.
Arrhythmias | From index CMR imaging to time of chart review, up to 5 years
  The number of patients with a diagnosis of an arrhythmia will be summarized and reported using basic descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Leandro Slipczuk, MD, PhD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Health System, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodriguez CJ, Allison M, Daviglus ML, Isasi CR, Keller C, Leira EC, Palaniappan L, Pina IL, Ramirez SM, Rodriguez B, Sims M; American Heart Association Council on Epidemiology and Prevention; American Heart Association Council on Clinical Cardiology; American Heart Association Council on Cardiovascular and Stroke Nursing. Status of cardiovascular disease and stroke in Hispanics/Latinos in the United States: a science advisory from the American Heart Association. Circulation. 2014 Aug 12;130(7):593-625. doi: 10.1161/CIR.0000000000000071. Epub 2014 Jul 14. PMID 25098323
- [Background] Daviglus ML, Talavera GA, Aviles-Santa ML, Allison M, Cai J, Criqui MH, Gellman M, Giachello AL, Gouskova N, Kaplan RC, LaVange L, Penedo F, Perreira K, Pirzada A, Schneiderman N, Wassertheil-Smoller S, Sorlie PD, Stamler J. Prevalence of major cardiovascular risk factors and cardiovascular diseases among Hispanic/Latino individuals of diverse backgrounds in the United States. JAMA. 2012 Nov 7;308(17):1775-84. doi: 10.1001/jama.2012.14517. PMID 23117778
- [Background] Barber S, Hickson DA, Wang X, Sims M, Nelson C, Diez-Roux AV. Neighborhood Disadvantage, Poor Social Conditions, and Cardiovascular Disease Incidence Among African American Adults in the Jackson Heart Study. Am J Public Health. 2016 Dec;106(12):2219-2226. doi: 10.2105/AJPH.2016.303471. Epub 2016 Oct 13. PMID 27736207
- [Background] Carnethon MR, Pu J, Howard G, Albert MA, Anderson CAM, Bertoni AG, Mujahid MS, Palaniappan L, Taylor HA Jr, Willis M, Yancy CW; American Heart Association Council on Epidemiology and Prevention; Council on Cardiovascular Disease in the Young; Council on Cardiovascular and Stroke Nursing; Council on Clinical Cardiology; Council on Functional Genomics and Translational Biology; and Stroke Council. Cardiovascular Health in African Americans: A Scientific Statement From the American Heart Association. Circulation. 2017 Nov 21;136(21):e393-e423. doi: 10.1161/CIR.0000000000000534. Epub 2017 Oct 23. PMID 29061565
- [Background] Hozawa A, Folsom AR, Sharrett AR, Chambless LE. Absolute and attributable risks of cardiovascular disease incidence in relation to optimal and borderline risk factors: comparison of African American with white subjects--Atherosclerosis Risk in Communities Study. Arch Intern Med. 2007 Mar 26;167(6):573-9. doi: 10.1001/archinte.167.6.573. PMID 17389288
- [Background] Patel AR, Kramer CM. Role of Cardiac Magnetic Resonance in the Diagnosis and Prognosis of Nonischemic Cardiomyopathy. JACC Cardiovasc Imaging. 2017 Oct;10(10 Pt A):1180-1193. doi: 10.1016/j.jcmg.2017.08.005. PMID 28982571
- [Background] Leiner T, Bogaert J, Friedrich MG, Mohiaddin R, Muthurangu V, Myerson S, Powell AJ, Raman SV, Pennell DJ. SCMR Position Paper (2020) on clinical indications for cardiovascular magnetic resonance. J Cardiovasc Magn Reson. 2020 Nov 9;22(1):76. doi: 10.1186/s12968-020-00682-4. PMID 33161900
- [Background] Romano S, Judd RM, Kim RJ, Heitner JF, Shah DJ, Shenoy C, Evans K, Romer B, Salazar P, Farzaneh-Far A. Feature-Tracking Global Longitudinal Strain Predicts Mortality in Patients With Preserved Ejection Fraction: A Multicenter Study. JACC Cardiovasc Imaging. 2020 Apr;13(4):940-947. doi: 10.1016/j.jcmg.2019.10.004. Epub 2019 Nov 11. PMID 31727563
- [Background] Puntmann VO, Carr-White G, Jabbour A, Yu CY, Gebker R, Kelle S, Hinojar R, Doltra A, Varma N, Child N, Rogers T, Suna G, Arroyo Ucar E, Goodman B, Khan S, Dabir D, Herrmann E, Zeiher AM, Nagel E; International T1 Multicentre CMR Outcome Study. T1-Mapping and Outcome in Nonischemic Cardiomyopathy: All-Cause Mortality and Heart Failure. JACC Cardiovasc Imaging. 2016 Jan;9(1):40-50. doi: 10.1016/j.jcmg.2015.12.001. PMID 26762873
- [Background] Kuruvilla S, Adenaw N, Katwal AB, Lipinski MJ, Kramer CM, Salerno M. Late gadolinium enhancement on cardiac magnetic resonance predicts adverse cardiovascular outcomes in nonischemic cardiomyopathy: a systematic review and meta-analysis. Circ Cardiovasc Imaging. 2014 Mar;7(2):250-258. doi: 10.1161/CIRCIMAGING.113.001144. Epub 2013 Dec 20. PMID 24363358
- [Background] Elliott P, Andersson B, Arbustini E, Bilinska Z, Cecchi F, Charron P, Dubourg O, Kuhl U, Maisch B, McKenna WJ, Monserrat L, Pankuweit S, Rapezzi C, Seferovic P, Tavazzi L, Keren A. Classification of the cardiomyopathies: a position statement from the European Society Of Cardiology Working Group on Myocardial and Pericardial Diseases. Eur Heart J. 2008 Jan;29(2):270-6. doi: 10.1093/eurheartj/ehm342. Epub 2007 Oct 4. PMID 17916581
- [Background] Maron BJ, Towbin JA, Thiene G, Antzelevitch C, Corrado D, Arnett D, Moss AJ, Seidman CE, Young JB; American Heart Association; Council on Clinical Cardiology, Heart Failure and Transplantation Committee; Quality of Care and Outcomes Research and Functional Genomics and Translational Biology Interdisciplinary Working Groups; Council on Epidemiology and Prevention. Contemporary definitions and classification of the cardiomyopathies: an American Heart Association Scientific Statement from the Council on Clinical Cardiology, Heart Failure and Transplantation Committee; Quality of Care and Outcomes Research and Functional Genomics and Translational Biology Interdisciplinary Working Groups; and Council on Epidemiology and Prevention. Circulation. 2006 Apr 11;113(14):1807-16. doi: 10.1161/CIRCULATIONAHA.106.174287. Epub 2006 Mar 27. PMID 16567565
- [Background] Rapezzi C, Arbustini E, Caforio AL, Charron P, Gimeno-Blanes J, Helio T, Linhart A, Mogensen J, Pinto Y, Ristic A, Seggewiss H, Sinagra G, Tavazzi L, Elliott PM. Diagnostic work-up in cardiomyopathies: bridging the gap between clinical phenotypes and final diagnosis. A position statement from the ESC Working Group on Myocardial and Pericardial Diseases. Eur Heart J. 2013 May;34(19):1448-58. doi: 10.1093/eurheartj/ehs397. Epub 2012 Dec 4. PMID 23211230